CLINICAL TRIAL: NCT03629834
Title: Internal and Predictive Validity of Epworth Sleepiness Scale to Evaluate Vigilance of Patient Treated for Obstructive Sleep Apnea Syndrome
Acronym: SAHOS-TIME
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2017_843_0034
Record Dates: First submitted 2018-07-16; First posted 2018-08-14 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Obstructive Sleep Apnea Syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Epworth Sleepiness Scale — Maintenance Wakefulness Test

SUMMARY:
Presently, there isn't any international recommendation to evaluate vigilance in Obstructive Sleep Apnea Syndrome. The French Society of Sleep Research and Medicine (SFRMS) recommend evaluating professional driver with a MWT but no recommendation exists for other patients. After a minimal treatment of 4 weeks, the physician has to evaluate the drowsiness risk of these patients using either an objective test like the MWT or a subjective one. In the university hospital Amiens-Picardie, since the 01/01/2015, every patient with an Obstructive Sleep Apnea Syndrome diagnosed by a polysomnography or a ventilatory polygraphy had a MWT after 4 weeks of treatment. At each time of the evaluation, Epworth Sleepiness Scale, tiredness score of Pichot, and depressive score of Beck are performed.

ELIGIBILITY:
Inclusion Criteria:

* patients treated by CPAP for Obstructive Sleep Apnea Syndrome

Exclusion Criteria:

* Central Apnea Syndrome
* Central Hypersomnia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: all patients more than 18 years treated by CPAP for Obstructive Sleep Apnea Syndrome diagnosed at the Sleep Medicine Unity of the Amiens Hospital having a MWT between the 01/01/15 and 31/12/16 were included. Patients were excluded if they had an Central Apnea Syndrome, Central Hypersomnia, no driving license or if they refused.
Sampling Method: Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2018-10-08 (Actual); Study Completion 2018-10-08 (Actual)

PRIMARY OUTCOMES:
Evaluation of the correlation between the MWT sleep latency scores and the results of the Epworth Sleepiness Scale after CPAP treatment | one day
  Three levels of vigilance are defined by the MWT : more than 34 min is rated as good vigilance; ≥ 20 et < 34 min as intermediate vigilance; under 20 min as bad vigilance.
Evaluation of the correlation between the MWT sleep latency scores and the results of the Epworth Sleepiness Scale after CPAP treatment | one day
  Two levels of vigilance are defined by the ESS score: score ≥11: bad vigilance, <11: good vigilance

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Basille D, Baud ME, Andrejak C, Basille-Fantinato A, Jounieaux V. Correlation between the Epworth Sleepiness Scale and the Maintenance of Wakefulness Test in Obstructive Sleep Apnea Patients Treated with Positive Airway Pressure. Respir Med Res. 2020 Nov;78:100787. doi: 10.1016/j.resmer.2020.100787. Epub 2020 Aug 28. PMID 32920453